CLINICAL TRIAL: NCT05982639
Title: Comparative Analysis of the Lung Inflammatory Response After Thoracic Surgery With Single or Double Lung Ventilation: a Randomized, Pilot, Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Felipe Dal Pizzol, Professor, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lung inflammation trial
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Thoracic Diseases; Surgery
MeSH Terms: conditions — Thoracic Diseases | interventions — One-Lung Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- one-lung ventilation (Other): Usual care. One lung ventilation will be provided using a Carleans type double lumen orotracheal tube.
  Interventions: Procedure: one lung ventilation
- two-lung ventilation and use of pneumothorax with CO2. (Experimental): Two lung ventilation will be provided using a single lumen orotracheal tube and CO2-induced pneumothorax
  Interventions: Procedure: two lung ventilation

INTERVENTIONS:
Procedure: two lung ventilation — The intervention do not involve a drug or device. It will be compared two different approaches to ventilate the lungs during the procedure . In this arm both lungs will be ventilated inserting a disposable trocar into the pleural cavity, and insufflating CO2 into the thoracic cavity via an insufflator. The insufflation pressure and the flow rate will be set as 8 mmHg and 10 l.min-1, of the cavity with CO2. The insufflator will be adjusted for cavity pressure in 8mmHg and flow of 10L/min.
  Arms: two-lung ventilation and use of pneumothorax with CO2.
Procedure: one lung ventilation — In this arm only one lung (the contralateral lung) will be ventilated using a Carlens type orotracheal tube
  Arms: one-lung ventilation

SUMMARY:
The goal of this clinical trial is to compare in patients undergoing thoracic procedures the lung inflammatory response in on one-lung ventilation and two-lung ventilation strategies The main question to answer is:

• Lung inflammation differs when comparing one to two-lung ventilation strategies during the procedure? Participants will be divided in the classic one lung ventilation or two lung ventilation (using pneumothorax with CO2) and different biomarkers of lung inflammation will be measured after procedures.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of pleural or mediastinal pathology that requires diagnostic or therapeutic surgical intervention;
* Written consent to participate

Exclusion Criteria:

* Pregnant women;
* Patients on mechanical ventilation prior to the procedure;
* Patients classified by the American Society of Anesthesiology (ASA) as class 4;
* Patients with subpulmonary or diaphragmatic pathologies, where it is believed that the two pulmonary technique is superior;
* Impossibility of using a double-lumen tube or difficult intubation;
* Patient does not support one-lung ventilation;
* Patient with previous lung resection surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Bronchoalveolar lavage fluid (BALF) levels of IL-6 | at a maximum 2 hours after the end of the thoracic procedure
  It will be compared the levels of IL-6 in the BALF collected immediately before and after the thoracic procedure

SECONDARY OUTCOMES:
Bronchoalveolar lavage fluid (BALF) levels of IL-8 | at a maximum 2 hours after the end of the thoracic procedure
  It will be compared the levels of IL-8 in the BALF collected immediately before and after the thoracic procedure
Bronchoalveolar lavage fluid (BALF) levels of IL-1 | at a maximum 2 hours after the end of the thoracic procedure
  It will be compared the levels of IL-1 in the BALF collected immediately before and after the thoracic procedure
Bronchoalveolar lavage fluid (BALF) levels of TNF | at a maximum 2 hours after the end of the thoracic procedure
  It will be compared the levels of TNF in the BALF collected immediately before and after the thoracic procedure
Bronchoalveolar lavage fluid (BALF) levels of oxidative stress | at a maximum 2 hours after the end of the thoracic procedure
  It will be compared the levels of malondialdehyde equivalents in the BALF collected immediately before and after the thoracic procedure
Post-procedure pulmonary complications | Until hospital discharge
  Composite outcome of associated pulmonary complications including pneumonia, re-expansion edema and postoperative non-re-expansion of the lung
Systemic levels of inflammatory and oxidative markers | at a maximum 2 hours after the end of the thoracic procedure
  Plasma levels of IL-6, IL-8, IL-1, TNF and malondialdehyde equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Balleter, MD, Principal Investigator — Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Locations (1):
- Hospital Azambuja, Brusque, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided